CLINICAL TRIAL: NCT03485872
Title: Urinary Incontinence Self-Screening for Healthy Aging
Brief Title: Urinary Incontinence Self-Screen for Healthy Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Retired Teachers of Ontario Foundation (Unknown); Interior Health (Industry)
Responsible Party: Principal Investigator, Kathy Rush, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: H17-03037
Record Dates: First submitted 2018-03-07; First posted 2018-04-02 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Screening and Referral Information (Experimental): The intervention will include a combination of self-screening and UI specific information and resources. Older adults in the intervention group will complete a gender specific UI Self-Screening tool. Men will complete the International Consultation on Incontinence Modular Questionnaire (ICIQ) for Males and women will complete the ICIQ for Females. In addition, the intervention group will receive a fact sheet with UI specific information, contact information to the local incontinence clinic and a link to a website with patient incontinence resources and education.
  Interventions: Other: Self-Screening and Referral Information
- Control Group (Active Comparator): Older adults assigned to the control group will receive standard care from their physicians. Standard care may differ from general practitioner to general practitioner. Usual care for urinary incontinence (UI) from general practitioners is generally minimal. Most patients do not tell their physicians about UI, and most physicians do not ask about UI. If this topic does come up during a GP appointment, a patient may be offered no treatment, lifestyle advice (e.g., do not drink before bed), told to do Kegels (but likely not instructed how to do these properly) or in some cases, offered pharmacological therapies (which will be captured in our questionnaire with the participants). But standard of care is unfortunately very often no care.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Self-Screening and Referral Information — Urinary incontinence self-screening questionnaire, fact sheet and self-referral information will be provided by mail or email.
  Arms: Self-Screening and Referral Information
Other: Standard Care — Demographic and quality of life questionnaires; standard care provided by participants' GPs
  Arms: Control Group

SUMMARY:
The purpose of this study is to increase awareness and timely treatment of urinary incontinence through a self-screening process. This is a 3 month study involving 2 activities; one taking place at the beginning of study and another 3 months later. Participants will be randomized into experimental and control groups. The experimental group will receive a demographic questionnaire, quality of life questionnaire, a questionnaire pertaining to urinary symptoms, information about how to self-screen for urinary incontinence and information regarding how to refer oneself to urinary incontinence resources. The control group will receive the demographic and quality of life questionnaires only. It is estimated that it will take participants 20-30 minutes to complete their package of questionnaires. After 3 months, the participants will receive a phone call inquiring into what actions they have taken regarding their urinary incontinence.

DETAILED DESCRIPTION:
Objectives: The overall aim is to increase awareness of urinary incontinence in community-based older adults and promote timely treatment. To achieve this aim the project objectives will include:

1. To develop a self-screening process for community-based older adults
2. To test the use of a self-screening process with community-based older adults

Methods:

Study Design: This study will use a pilot randomized control trial to test the effectiveness of a self-screening process with older adults. The hypothesis is that older adults exposed to the self-screening process will follow up with health professionals to receive help for the UI condition. There will be two groups of older adults. The intervention group will participate in self-screening and the control will not be exposed to self-screening. Using this approach is necessary to determine whether or not the self-screening works.

Setting: Senior's Centers and organizations dedicated to seniors in Kelowna, West Kelowna and Lake Country will serve as the recruitment sites for this study. These Senior's Centers/organizations (e.g., Lake Country Seniors Centre, Lake Country Health Planning Society, Westside Health Network, Seniors Outreach Bureau) serve large and different populations of seniors (>300 seniors) so overlap in membership is not expected to be an issue. Excel randomization function will be used to assign participants to one of the two arms (the arm receiving the self-screening process or the arm not receiving this process). The randomization assignments (allocations) will be placed in individual sealed envelopes. After informed consent is obtained, the Research Assistant (RA) will choose the next available envelope to reveal which arm the study participant will be assigned.

Data Collection:

Pre-test: Prior to implementation, the self-screening tool will be pre-tested with 5 older adults attending participating seniors centres/organizations. The purpose of the pretest will be to identify any implementation issues such as recruitment, administration, understanding and ease of use of the self-screening tools.

Procedures: Older adults assigned to both groups will receive follow up from the RA who will provide details about the study and answer any questions. Prior to randomization, consenting older adults from both groups will complete a demographic (e.g., age, sex, highest level of education, household income), health history profile (e.g., co-morbidities, history of previous referrals for UI, medications) (see Demographic and Health History Profile) and a quality of life questionnaire 17 (see The King's Health Questionnaire).

Three months following study entry participants from both groups will receive a phone follow-up to obtain information about actions they have taken re IU (e.g., self/physician referral), UI symptoms, treatments received, satisfaction with care, and changes in quality of life. The follow up phone call will be recorded. It is expected the baseline and 3 month follow up data collection will take approximately 20-30 minutes to complete.

Post-Intervention Focus Groups: To obtain feedback on the self-screening process, focus groups (n=2) will be conducted with older adults (10-12 participants) who were in the self-screening group. At the end of 3-months from study entry, in conjunction with survey completion, participants will be invited to participate in a focus group. Those expressing an interest in focus group participation will be contacted with details of the date, time of the focus group and will receive a copy of the semi-structured interview questions. Questions will address participants' comfort with the self-screening process, rationale and influences on choice to self-refer or not, barriers/facilitators to self-referral, recommendations to make the self-screening process easier.

Data Analysis: Analysis will include a description of sample and primary and secondary analyses.

Description of Sample:

Frequency analysis will be conducted on all demographic (age, sex, highest level of education, household income), health history profile (co-morbidities, history of previous referrals for UI, medications) and quality of life. For continuous variables, means with associated standard deviations (SD) will be calculated for parametric variables or medians with associated interquartile ranges will be calculated for nonparametric variables. For categorical variables, percentages with 95% confidence interval (CI) will be calculated. These calculations will be calculated for the total study population as well as for participants in each study group.

Primary analysis:

The study hypothesis is that older adults exposed to the self-screening process will follow-up with health professionals to receive help for their UI condition more often than the control group. To test this hypothesis investigators will calculate the proportion (with 95% CI) of participants who self-report as having self-referred to a health professional (binary yes/no response) during the study period for each group. A chi-square test will be conducted to determine if the self-screening process is associated with self-referral to a health professional. In addition, a logistic regression analysis will be conducted to model the odds of self-referring among participants who have undergone self-screening, adjusting for demographics, and health history variables. Bivariate analysis will be conducted and variables significantly associated with self-referral will be entered into the model. Since the sample size will only allow for having 3 variables in the model, more than one regression model may be necessary. If this is the case, a Bonferroni adjustment will be used to account for multiple comparisons.

Secondary analysis:

Quality of life scores will be compared within and between groups. For the within group comparison, a two-sided dependent t-test will be conducted using the pre study and 3-month quality of life scores for each group. To determine if a change in quality of life (difference between pre study and 3-mont quality of life scores) is statistically significant and mixed between-within subjects analysis of variance will be conducted.

All participants will complete a Urinary Symptoms questionnaire (ICIQ-FLUTS) which consists of ordinal categorical responses to questions related to urinary symptoms. Each question has five response options. For each question, each response category will be assigned a numeric value depending on the severity of the symptom (1= no symptoms; 5=severe symptoms). For each participant, improvement in symptoms will be determined by a reduction in the ordinal value. Improvement in UI symptoms will be compared between groups using a chi-square test.

Investigators are also interested in knowing if self-screening results in higher proportion of participants initiating medication of UI during the study period. Therefore, the proportion of participants in each group who started medication for UI during the study period will be compared using a chi-square test.

Limitations: It is possible that screening for eligibility for the study may make a person more likely to self-refer. If this occurs in the control arm, it may bias the results toward the null hypothesis (i.e. it may be less likely to detect a difference between study arms).

ELIGIBILITY:
Inclusion Criteria:

* Adults 65 years of age and older
* Attend a local Senior's Centre or organization
* Report having some UI symptoms
* Living independently
* Ambulatory
* No more than mild cognitive impairment
* Able to read and write in English or have someone who can assist with reading the data collection information and can complete a paper survey independently

Exclusion Criteria:

* Cognitive impairment
* Require more than minimal assistance with completing the survey
* Any impairment (e.g., vision) that would make self-screening and follow up challenging.
* Have been referred to a UI specialist or continence program in the past

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Self-Referral Questionnaire | 3 months
  The primary outcome will be the number of older adults who take action to receive help for their UI. The following question will be asked through a questionnaire at three month follow-up: "During the past three months, what have you done about the leakage?" Participants will have the option to check off any of the following options: "I haven't done anything about it", "have seen my GP about it", and "referred myself to the local Urinary Incontinence Clinic".

SECONDARY OUTCOMES:
Treatments Received Questionnaire | 3 months
  The treatments the participants receive as a result of self-referral for their urinary incontinence will be noted. The following question will be asked through a questionnaire at three month follow-up: "What treatments have you received?" Participants will have the option to check off any of the following options: Lifestyle treatments/education by a health care practitioner (ex. fluid management, kegel exercises, etc.)"; "prescription medication treatments"; and "surgical treatments".
Satisfaction with Care Questionnaire | 3 months
  Participants' satisfaction with the care they receive will be observed, factoring in whether or not they received the intervention. The following question will be asked through a questionnaire at three month follow-up: "How satisfied have you been with the care you have been receiving for urinary incontinence?" Participants will have the option to check off one of the following options: "poor", "fair", "good", "very good", or "excellent".

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Rush, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donovan JL, Abrams P, Peters TJ, Kay HE, Reynard J, Chapple C, De La Rosette JJ, Kondo A. The ICS-'BPH' Study: the psychometric validity and reliability of the ICSmale questionnaire. Br J Urol. 1996 Apr;77(4):554-62. doi: 10.1046/j.1464-410x.1996.93013.x. PMID 8777617
- [Background] Jackson S, Donovan J, Brookes S, Eckford S, Swithinbank L, Abrams P. The Bristol Female Lower Urinary Tract Symptoms questionnaire: development and psychometric testing. Br J Urol. 1996 Jun;77(6):805-12. doi: 10.1046/j.1464-410x.1996.00186.x. PMID 8705212
- [Background] Okamura K, Nojiri Y, Osuga Y. Reliability and validity of the King's Health Questionnaire for lower urinary tract symptoms in both genders. BJU Int. 2009 Jun;103(12):1673-8. doi: 10.1111/j.1464-410X.2008.08335.x. Epub 2009 Jan 9. PMID 19154505

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03485872/Prot_SAP_001.pdf